CLINICAL TRIAL: NCT04661072
Title: Congenital Uterine Anomalies: Identifying Cancer Associations and Genetic and Environmental Factors to Improve Clinical Care
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000028592; 1R03HD109641-01A1 (NIH)
Record Dates: First submitted 2020-12-08; First posted 2020-12-09 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Congenital Uterine Anomaly
Keywords: Cancer associations; Environmental factors
MeSH Terms: conditions — Uterine Anomalies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Following informed consent, blood will be collected for genetic evaluation. DNA will be extracted from EDTA-blood and analyzed using an integrated approach of microarray for copy number variations (CNV), and Whole Exome Sequencing (WES) for Single Nucleotide Variation (SNV).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Congenital Uterine Anomalies (CUA): The rates of renal, breast, uterine, ovarian and vaginal cancers in women who have been diagnosed with a CUA will be studies

SUMMARY:
The purpose of this research study is to learn more about the health outcomes associated with congenital uterine anomalies (CUAs), and the possible environmental and genetic causes of the condition. The researchers plan to investigate whether any cancer associations (with breast, renal, ovarian, vaginal and uterine cancers) exist in females with CUAs. The investigator will also investigate any environmental and genetic factors that may be responsible for causing CUAs.

DETAILED DESCRIPTION:
Aim 1: To identify female subjects diagnosed with a Congenital Uterine Anomaly (CUA) receiving care at Yale New Haven Health.

Aim 2: Identify (i) the prevalence of renal, breast, ovarian, uterine and vaginal cancers associated with CUAs, and (ii) the association of environmental factors, via a survey obtained by phone, email or interview.

Aim 3: Conduct genetic evaluation of the index subjects, parents, sister(s) (as feasible), and female offspring to identify potential causes and patterns of inheritance using whole exome sequencing (WES) and microarray.

Following informed consent, blood will be collected for genetic evaluation. DNA will be extracted from EDTA-blood and analyzed using an integrated approach of microarray for copy number variations (CNV), and Whole Exome Sequencing (WES) for Single Nucleotide Variation (SNV).

Undertaking review of the medical records will identify the cohort of patients we wish to survey to then ascertain further information regarding their CUA diagnosis and other related details. The information to be elicited from the survey are outlined in the attached survey questions. Key associations we seek to investigate include (1) the type and prevalence of renal, breast, ovarian, uterine and vaginal cancers among patients with Mullerian Anomaly, and (2) identifying potential in-utero exposure to particular environmental agents in patients with CUAs.

Review of the medical records will enable us to undertake this first key step of establishing a cohort of subjects with MA and an initial data set related to their specific health information. We anticipate further investigations may build upon this initial data set, both with the cohort established, and more broadly with collaborators and additional national and international cohorts of patients with MA.

ELIGIBILITY:
Inclusion Criteria:

* females
* age: 13 or older
* encounters limited to: Yale New Haven Hospital, Bridgeport Hospital, Greenwich Hospital and Lawrence+ Memorial Hospital.
* diagnosis of any variation of CUA

Exclusion Criteria:

* who will decline to participate in a study upon contact
* non-English speaking except Spanish speaking
* unable to participate in consent or assent process due to mental disability

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women and girls who have received care within the Yale New Haven Health system and have a CUA diagnosis Anticipated number - approximately 300 subjects Age range - from 13 years old and older Health status - able to participate in consent and assent (based on age) process
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of breast cancer in women with CUA's compared to women without CUA's | 6-months
  Prevalence of breast cancer in women with CUA's compared to women without CUA's will be measured
Prevalence of ovarian cancer in women with CUA's compared to women without CUA's | 6-months
  Prevalence of ovarian cancer in women with CUA's compared to women without CUA's will be measured
Prevalence of uterine cancer in women with CUA's compared to women without CUA's | 6-months
  Prevalence of uterine cancer in women with CUA's compared to women without CUA's will be measured
Prevalence of cervical cancer in women with CUA's compared to women without CUA's | 6 month
  Prevalence of cervical cancer in women with CUA's compared to women without CUA's will be measured
Prevalence of vaginal cancer in women with CUA's compared to women without CUA's | 6 month
  Prevalence of vaginal cancer in women with CUA's compared to women without CUA's will be measured
Prevalence of renal cancer in women with CUA's compared to women without CUA's | 6 month
  Prevalence of renal cancer in women with CUA's compared to women without CUA's will be measured

SECONDARY OUTCOMES:
Whole exome sequencing (WES) and microarray | 24 months
  WES and microarray will be conducted in subjects with CUAs. The discovery of possible causative genes would be measured using yes/no outcome variable.

CONTACTS AND LOCATIONS:
Overall Officials: Alla Vash-Margita, MD, Principal Investigator — Yale University; Emanuele Pelosi, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States